CLINICAL TRIAL: NCT05308329
Title: Kitasato Percutaneous Coronary Intervention Registry
Brief Title: Kitasato PCI Registry
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kitasato University (Other)
Responsible Party: Principal Investigator, Yoshiyasu Minami, Assistant Professor, Kitasato University
Other Study IDs: KITASATO-B18-099
Record Dates: First submitted 2022-01-11; First posted 2022-04-04 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Acute Coronary Syndrome; STEMI - ST-segment Elevation Myocardial Infarction; NSTEMI - Non-ST-Segment Elevation Myocardial Infarction; Atherosclerosis; Coronary; Ischemic; Stable Angina
MeSH Terms: conditions — Acute Coronary Syndrome; Atherosclerosis; Ischemia; Angina, Stable

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Intra-coronary imaging device — Culprit/nonculprit lesions are accessed by intra-coronary imaging device including intravascular ultrasound and optical coherence tomography.
Behavioral: PCI procedural characteristics — Procedural characteristics include the information about angiographical characteristics, type of stent, pre/post POBA, and thrombectomy.

SUMMARY:
The Kitasato PCI Registry is a single-center, observational, prospective study. This study aims to investigate the impact of characteristics in clinical manifestation, patients' background, procedure of percutaneous coronary intervention (PCI), and pre/post PCI culprit/nonculprit lesion observed by intra-coronary imaging modality on clinical outcomes.

DETAILED DESCRIPTION:
Subjects who underwent PCI are eligible in this registry. The analysis for clinical characteristics, PCI procedural characteristics and findings of intra-coronary imaging including optical coherence tomography (OCT) and intravascular ultrasound (IVUS) is conducted. Subjects are clinically followed up to 5 years after the PCI.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent PCI

Exclusion Criteria:

* Patients who did not agree to participate in the registry

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with coronary artery disease requiring PCI at Kitasato University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 4500 (Estimated)
Dates: Start 2012-02-01 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Device-oriented clinical end points (DoCE) | 5 years after the PCI
  Composite of all-cause death, myocardial infarction, ischemic stroke, clinically indicated Composite of cardiac death, target lesion revascularization and stent thrombosis

SECONDARY OUTCOMES:
Major adverse cardiac and cerebrovascular events (MACCE) | 5 years after the PCI
  Composite of all-cause death, myocardial infarction, ischemic stroke, clinically indicated coronary revascularization

CONTACTS AND LOCATIONS:
Overall Officials: Yoshiyasu Minami, Principal Investigator — Kitasato University School of Medicine
Locations (1):
- Kitasato University Hospital, Sagamihara, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Asakura K, Minami Y, Kinoshita D, Katamine M, Kato A, Katsura A, Sato T, Muramatsu Y, Hashimoto T, Kameda R, Meguro K, Shimohama T, Ako J. Impact of triglyceride levels on plaque characteristics in patients with coronary artery disease. Int J Cardiol. 2022 Feb 1;348:134-139. doi: 10.1016/j.ijcard.2021.12.008. Epub 2021 Dec 9. PMID 34896410
- [Background] Kato A, Minami Y, Asakura K, Katamine M, Katsura A, Muramatsu Y, Sato T, Kakizaki R, Hashimoto T, Meguro K, Shimohama T, Ako J. Characteristics of carotid atherosclerosis in patients with plaque erosion. J Thromb Thrombolysis. 2021 Aug;52(2):620-627. doi: 10.1007/s11239-021-02419-1. Epub 2021 Mar 10. PMID 33694096
- [Background] Hashimoto T, Minami Y, Asakura K, Katamine M, Kato A, Katsura A, Sato T, Muramatsu Y, Kakizaki R, Fujiyoshi K, Ishida K, Kameda R, Meguro K, Shimohama T, Ako J. Achilles tendon thickening is associated with higher incidence of adverse cardiovascular event in patients with coronary artery disease. Heart Vessels. 2021 Feb;36(2):163-169. doi: 10.1007/s00380-020-01679-w. Epub 2020 Aug 6. PMID 32761364
- [Background] Muramatsu Y, Minami Y, Kato A, Katsura A, Sato T, Kakizaki R, Nemoto T, Hashimoto T, Fujiyoshi K, Meguro K, Shimohama T, Ako J. Lipoprotein (a) level is associated with plaque vulnerability in patients with coronary artery disease: An optical coherence tomography study. Int J Cardiol Heart Vasc. 2019 Jun 13;24:100382. doi: 10.1016/j.ijcha.2019.100382. eCollection 2019 Sep. PMID 31245530
- [Background] Kakizaki R, Minami Y, Hashikata T, Nemoto T, Hashimoto T, Fujiyoshi K, Meguro K, Shimohama T, Tojo T, Ako J. Impact of underlying plaque type on strut coverage in the early phase after drug-eluting stent implantation. Coron Artery Dis. 2018 Dec;29(8):624-631. doi: 10.1097/MCA.0000000000000654. PMID 29975201
- [Background] Kakizaki R, Minami Y, Katamine M, Katsura A, Muramatsu Y, Hashimoto T, Meguro K, Shimohama T, Ako J. Clinical outcome of biodegradable polymer sirolimus-eluting stent and durable polymer everolimus-eluting stent in patients with diabetes. Cardiovasc Diabetol. 2020 Oct 1;19(1):162. doi: 10.1186/s12933-020-01145-x. PMID 33004019
- [Background] Fujiyoshi K, Minami Y, Ishida K, Kato A, Katsura A, Muramatsu Y, Sato T, Kakizaki R, Nemoto T, Hashimoto T, Sato N, Meguro K, Shimohama T, Tojo T, Ako J. Incidence, factors, and clinical significance of cholesterol crystals in coronary plaque: An optical coherence tomography study. Atherosclerosis. 2019 Apr;283:79-84. doi: 10.1016/j.atherosclerosis.2019.02.009. Epub 2019 Feb 14. PMID 30802681